CLINICAL TRIAL: NCT03148392
Title: A Prospective Comparison of Quality of Life Following Atrial Fibrillation Ablation Using the Arctic Front Advance Cryo Balloon Compared to Contact Force Sensing Radiofrequency Catheter Ablation
Brief Title: Assess Differences in Pain Following Cryo and Radiofrequency Atrial Fibrillation Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sumit Verma, MD (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Sumit Verma, MD, Principal Investigator, Langhorne Cardiology Consultants, Inc.
Organization: Langhorne Cardiology Consultants, Inc. (Other)
Other Study IDs: Cryo RF Ablation QOL
Record Dates: First submitted 2017-04-27; First posted 2017-05-11 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Cryo Balloon Ablation: Arctic Front Advance Cryo Balloon: Mode of ablation determined based on patient and physician preference
- Radiofrequency Ablation: Contact Force Sensing Radiofrequency Catheter Ablation: Mode of ablation determined based on patient and physician preference

SUMMARY:
The primary objective is to assess any differences in patient quality of life between Cryo Balloon ablation and Radiofrequency ablation in the treatment of atrial fibrillation. The study will also assess any differences in the amount and duration of pain medication required after the ablation.

DETAILED DESCRIPTION:
Currently there are several different accepted techniques for performing ablation of atrial fibrillation. The two primary techniques currently in use in our center for atrial fibrillation are Cryo Balloon and Radiofrequency ablation.

Based on personal observation, it is felt that patients undergoing Radiofrequency ablation have a higher incidence of chest discomfort and subsequently a greater requirement for pain medications post procedure as compared to those patients undergoing Cryo ablation.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation who are advised either Cryoablation or Radiofrequency ablation for treatment.

Exclusion Criteria:

* Persistent atrial fibrillation
* Pregnant
* Taking pain medications for acute or chronic conditions at the time of the procedure.
* Undergo a combination of Cryoablation and Radiofrequency ablation
* Radiofrequency group who undergo ablation beyond pulmonary vein isolation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measurement | 7 Days
  Self report pain intensity measured at baseline and then once a day beginning at least four hours after the ablation. Three individual pain scales will be used. Universal Pain Assessment Tool is scored 0 to 10 with 0 = no pain and 10 = severe.

SECONDARY OUTCOMES:
Health Status and Activity Measurement | 7 Days
  Self report health status and activity measured at baseline and then once a day beginning at least four hours after the ablation using SF-36 Health and Well-Being Questionnaire.
Pain Medication Assessment | 30 Days
  Assess amount and duration of pain medication required post ablation

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Verma, MD, Principal Investigator — Cardiology Consultants
Locations (1):
- Cardiology Consultants, Pensacola, Florida, United States

IPD SHARING:
Plan to Share IPD: No